CLINICAL TRIAL: NCT06592664
Title: A Phase 1b/2a, Double-blind, Placebo-controlled, Three Arm, Randomized Study Evaluating a Single Intravenous Push Followed by a Continuous Infusion of Certepetide Over 4 Hours When Added to Standard of Care (SoC) Versus Two Intravenous Pushes of Certepetide When Added to SoC, Versus SoC Alone in Subjects With Previously Untreated Metastatic Pancreatic Ductal Adenocarcinoma (FORTIFIDE)
Brief Title: Certepetide Phase 1b/2a Continuous Infusion Trial in mPDAC
Acronym: FORTIFIDE
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Management Decision
Sponsor: Lisata Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LSTA1-P06
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Pancreas Cancer; Pancreatic Carcinoma; Pancreas Adenocarcinoma; Pancreatic Ductal Adenocarcinoma; Unresectable Pancreatic Cancer; Metastatic Pancreatic Cancer; PDAC; PDAC - Pancreatic Ductal Adenocarcinoma
Keywords: Chemo; Chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SoC chemotherapy plus one certepetide IV push, one placebo IV push, and certepetide infusion (Experimental)
  Interventions: Drug: certepetide; Drug: nab-paclitaxel; Drug: gemcitabine; Drug: placebo matching certepetide
- SoC chemotherapy plus two certepetide IV pushes and placebo infusion (Experimental)
  Interventions: Drug: nab-paclitaxel; Drug: gemcitabine; Drug: certepetide; Drug: placebo matching certepetide
- SoC chemotherapy plus two placebo IV pushes and placebo infusion (Active Comparator)
  Interventions: Drug: nab-paclitaxel; Drug: gemcitabine; Drug: placebo matching certepetide

INTERVENTIONS:
Drug: certepetide — certepetide given as an IV push over 1 minute and as an IV infusion over 4 hours when standard treatment(s) are given
  Other Names: LSTA1; CEND-1
  Arms: SoC chemotherapy plus one certepetide IV push, one placebo IV push, and certepetide infusion
Drug: nab-paclitaxel — nab-paclitaxel 125 mg/m^2 IV administered on Day 1, 8, and 15 every 28 days
  Other Names: Abraxane
Drug: gemcitabine — gemcitabine 1000 mg/m^2 IV administered on Day 1, 8, and 15 every 28 days
Drug: placebo matching certepetide — placebo given as two IV pushes over 1 minute and as an IV infusion over 4 hours when standard treatment(s) are given
  Arms: SoC chemotherapy plus two placebo IV pushes and placebo infusion
Drug: certepetide — certepetide given as two IV pushes over 1 minute when standard treatment(s) are given
  Other Names: LSTA1; CEND-1
  Arms: SoC chemotherapy plus two certepetide IV pushes and placebo infusion
Drug: placebo matching certepetide — placebo given as an IV infusion over 4 hours when standard treatment(s) are given
  Arms: SoC chemotherapy plus two certepetide IV pushes and placebo infusion
Drug: placebo matching certepetide — certepetide given as a slow IV push over 1 minute when standard treatment(s) are given
  Arms: SoC chemotherapy plus one certepetide IV push, one placebo IV push, and certepetide infusion

SUMMARY:
The goal of this clinical trial is to test a new drug plus standard treatment compared with standard treatment alone in people with metastatic pancreatic ductal adenocarcinoma.

The main questions it aims to answer are:

* is the new drug plus standard treatment safe and tolerable
* is the new drug plus standard treatment more effective than standard treatment

Participants will:

* Visit the clinic three times every 28 days for treatment and tests
* Have CT or MRI scans every 8 weeks while on treatment

DETAILED DESCRIPTION:
This is a Phase 1b/2a, double-blind, placebo-controlled, three-arm, randomized study evaluating a single intravenous push of certepetide followed by a continuous infusion of certepetide over 4 hours when added to standard of care (SoC) versus two intravenous pushes of certepetide given 4 hours apart when added to SoC, versus SoC alone in people with previously untreated metastatic pancreatic ductal adenocarcinoma (mPDAC).

The study will consist of a screening period, a run-in period, a treatment period, an end-of-treatment follow-up visit, and a long-term follow up period.

Participants who provide informed consent will be screened for eligibility within 28 days prior to beginning the study treatment run-in period. Once eligibility is confirmed, participants will be randomized to one of the three treatment groups.

During the 3-day run-in period, participants will only receive the LSTA1 or placebo components of their randomized treatment regimen. After the 3-day run-in, Cycle 1 of treatment will commence. Tumor scans will be performed every 8 weeks (56 days ± 7 days) while on treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic pancreatic ductal adenocarcinoma that has not been treated previously and be eligible for treatment with nab-paclitaxel and gemcitabine
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy ≥ 3 months
* At least one measurable tumor lesion as assessed by RECIST 1.1
* Adequate organ and marrow function
* Adequate contraception

Exclusion Criteria:

* Concurrent use of any other anti-cancer therapy including chemotherapy, targeted therapy, immunotherapy, or biological agents
* Received prior anti-cancer therapy for their pancreatic cancer
* Any condition or comorbidity that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of subject safety or study results, including but not limited to:

  * Any major surgery or irradiation less than 4 weeks prior to baseline disease assessment
  * Active infection (viral, fungal, or bacterial) requiring systemic therapy
  * Known active hepatitis B virus, hepatitis C virus, or HIV infection
  * Active tuberculosis as defined per local guidance
  * History of allogeneic tissue/solid organ transplant
  * Prior malignancy requiring active treatment within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast
  * Pregnant or breastfeeding
  * Clinically significant or symptomatic cardiovascular/cerebrovascular disease (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) within 6 months before randomization
* History or clinical evidence of symptomatic central nervous system (CNS) metastases
* Enrolled in any other clinical protocol or investigational trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2030-01 (Estimated); Primary Completion 2035-01 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | 30 days after treatment discontinuation
  The National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE) will be used to grade the intensity of adverse events throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Kristen K. Buck, MD, Study Chair — Lisata Therapeutics, Inc.

IPD SHARING:
Plan to Share IPD: No